CLINICAL TRIAL: NCT02895412
Title: A Clinical Trial of Donor-derived WT1 Specific T Cells for Prevention of Relapse in Combination With Multiple Pathogen Specific T Cells for Prevention of Infection in Patients Undergoing Allogeneic Haemopoietic Stem Cell Transplant for AML
Brief Title: Infection and Tumour Antigen Cellular Therapy
Acronym: INTACT-WT1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sydney (Other)
Responsible Party: Principal Investigator, Dr Emily Blyth, Dr, University of Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: INTACT-WT1
Record Dates: First submitted 2016-02-23; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Leukemia, Myelocytic, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplant Recipient (Experimental): The T cell product administration is personalized cellular therapy product, individually prepared for each participant.
  Donor-derived WT1-CTL and P-CTL.
  It's exact make up and effect is dependent on both donor and recipient characteristics and as such variability is expected in the response. These variations will be adjusted for by multiple samplings over time and collation and analysis of response in both individuals an the group as a whole.
  One infusion of 2 x 107/m2 P-CTLs prophylactically on or after day 28 post-allogeneic peripheral blood haemopoietic stem cell transplant (HSCT), combined with up to four infusions of 2x107/m2 WT1-CTLs.
  Interventions: Biological: Donor-derived WT1-CTL and P-CTL

INTERVENTIONS:
Biological: Donor-derived WT1-CTL and P-CTL — Donor-derived WT1-CTL and P-CTL.
  P-CTL will be given prophylactically a minimum of 28 days after transplantation followed by administration of monthly infusions of WT1-CTL for up to four doses.

SUMMARY:
This study is to test a new therapy for patients with acute myeloid leukaemia who are undergoing blood stem cell transplant. In this study, the investigators will take a small number of your immune cells whose normal function is to give immunity to infections and help to fight leukaemia. These cells will be stimulated to multiply in the laboratory and will then be given to the transplant recipient after the transplant. This is a sort of "immunity transplant". The exact purpose of this study is to investigate if these cells are safe and effective in patients having a transplant for AML.

DETAILED DESCRIPTION:
The study will analyse the safety and biological efficacy of administering the investigational products (donor-derived Wilm's Tumour Antigen-specific cytotoxic T lymphocytes and with cytotoxic T lymphocytes specific for multiple opportunistic pathogens (cytomegalovirus (CMV), Adenovirus (Adv), Epstein Barr virus (EBV), Varicella-Zoster virus (VZV), Influenza, BK virus (BKV), and fungal infections), hereafter referred to as P-CTLs) for the prophylaxis of relapse, viral and fungal reactivation and infection following allogeneic blood or marrow transplantation for acute myeloid leukaemia. P-CTL will be given prophylactically a minimum of 28 days after transplantation followed by administration of monthly infusions of WT1-CTL for up to four doses. Our aims are to study the safety of combining WT1-CTL and P-CTL infusions; their persistence, effect on relapse of disease, effect on minimal residual disease, reconstitution of WT-1 and pathogen-specific immunity, viral reactivation, infection rates after transplantation, viral load; use of antiviral and antifungal pharmacotherapy for specific infections, hospitalisations and overall survival. Safety of infusions with respect to the development of adverse events within the first 12 months post-transplant will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing myeloablative or non-myeloablative allogeneic transplantation from an HLA (A, B and DR) identical or 1-3 antigen mismatched family or unrelated donor
2. Transplant performed for acute myeloid leukaemia
3. Leukaemia blasts express the WT1 tumour antigen as determined by the European LeukaemiaNet standardised assay described in 16. WT1 overexpression will be defined by greater than 250 copies/104ABL copies in bone marrow samples or greater than 50 copies/104ABL copies in peripheral blood. This assay will be performed on samples collected as part of routine clinical care at diagnosis and during initial treatment prior to transplantation. Testing will be performed after consent for trial participation has been obtained and negativity for WT1 will be classified as screening failure
4. Recipients of peripheral blood HSCT
5. Adequate hepatic and renal function (< 3 x upper limit of normal for AST, ALT, < 2 x upper limit of normal for total bilirubin, serum creatinine)
6. Estimated life expectancy of at least 12 months
7. Patient (or legal representative) has given informed consent

Exclusion Criteria:

1. Use of anti-lymphocyte globulin (ALG, ATG, Campath or other broad spectrum lymphocyte antibody) given in the 4 weeks immediately prior to infusion or planned within 4 weeks after infusion
2. Grade II or greater graft versus host disease within 1 week prior to infusion
3. Prednisone or methylprednisone at a dose of > 1 mg/kg (or equivalent in other steroid preparations) administered within 72 hours prior to cell infusion
4. Prior allogeneic HSCT
5. Privately insured in or outpatients (see Indemnity Issues, Section 11.4)

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 Years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Hospital, Westmead, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No